CLINICAL TRIAL: NCT02646826
Title: Paxerol™ (a Novel Formulation of Acetaminophen and Ibuprofen) for Treatment of Nocturia - A Phase II Placebo-Controlled Trial
Brief Title: Paxerol™ for Treatment of Nocturia - A Phase II Placebo-Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wellesley Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-Paxerol-002
Record Dates: First submitted 2015-12-30; First posted 2016-01-06 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Subjects are treated with placebo tablets.
  Interventions: Other: Placebo
- Paxerol - Dose Level 1 (Experimental): Subjects are treated with the first dose level of Paxerol.
  Interventions: Drug: Paxerol - Dose Level 1
- Paxerol - Dose Level 2 (Experimental): Subjects are treated with the second dose level of Paxerol.
  Interventions: Drug: Paxerol - Dose Level 2
- Paxerol - Dose Level 3 (Experimental): Subjects are treated with the third dose level of Paxerol.
  Interventions: Drug: Paxerol - Dose Level 3

INTERVENTIONS:
Other: Placebo — Subjects are treated with Placebo tablets
  Other Names: Placebo control
  Arms: Placebo
Drug: Paxerol - Dose Level 1 — Subjects are treated with the first dose level of Paxerol
  Other Names: Treatment arm 1
  Arms: Paxerol - Dose Level 1
Drug: Paxerol - Dose Level 2 — Subjects are treated with the second dose level of Paxerol
  Other Names: Treatment arm 2
  Arms: Paxerol - Dose Level 2
Drug: Paxerol - Dose Level 3 — Subjects are treated with the third dose level of Paxerol
  Other Names: Treatment arm 3
  Arms: Paxerol - Dose Level 3

SUMMARY:
This is a multi-center, double-blind, placebo-controlled study with two weeks of daily oral administration of one of three dose levels of Paxerol or placebo in subjects with nocturia. Eligible study subjects will be identified according to inclusion/exclusion criteria (see below), and baseline assessments will be recorded.

Due to small sample size of 25 patients per group in this proof-of-principle dosing-finding trial, stratification according to gender and BMI will be difficult. However, similar distribution of patient types to the four treatment groups will be attempted by evenly assigning patients to the four treatment groups according to genders and body mass index (BMI) of <25, 25-30 and 30-40.

Paxerol or placebo will be taken 30 minutes before bedtime daily for two weeks. Nocturia frequency, Nocturia Quality of Life (NQOL), Duration of First Undisturbed Sleep (DFUS), total hours of nightly sleep, safety and tolerability will be monitored before and after a two-week treatment period. Results from subjects treated with different doses of Paxerol and placebo will be assessed and compared. Baseline urinary Prostaglandin E2 (PGE2) production will also be assayed to assess potential correlation between baseline urinary PGE2 production and responsiveness to Paxerol treatment.

DETAILED DESCRIPTION:
The co-primary objectives are:

A. To assess the effect of different doses of Paxerol on the reduction in the number of nocturia episodes.

B. To assess the clinical benefit of different doses of Paxerol in reducing nocturia via assessment of nocturia quality of life (NQOL).

The secondary objectives are to assess the effects of different doses of Paxerol on:

A. Duration of First Undisturbed Sleep (DFUS) B. Total hours of nightly sleep C. Safety and tolerability

An exploratory assessment is to evaluate baseline urinary PGE2 production on the responsiveness of subjects to Paxerol.

This is a multi-center, double-blind, placebo-controlled study with two weeks of daily oral administration of one of three dose levels of Paxerol or placebo in subjects with nocturia. Eligible study subjects will be identified according to inclusion/exclusion criteria (see below), and baseline assessments will be recorded.

Due to small sample size of 25 patients per group in this proof-of-principle dosing-finding trial, stratification according to gender and BMI will be difficult. However, similar distribution of patient types to the four treatment groups will be attempted by evenly assigning patients to the four treatment groups according to genders and body mass index (BMI) of <25, 25-30 and 30-40.

Paxerol or placebo will be taken 30 minutes before bedtime daily for two weeks. Nocturia frequency, Nocturia Quality of Life (NQOL), Duration of First Undisturbed Sleep (DFUS), total hours of nightly sleep, safety and tolerability will be monitored before and after a two-week treatment period. Results from subjects treated with different doses of Paxerol and placebo will be assessed and compared. Baseline urinary Prostaglandin E2 (PGE2) production will also be assayed to assess potential correlation between baseline urinary PGE2 production and responsiveness to Paxerol treatment.

Study duration for each subject is approximately 4 weeks, which includes screening, baseline assessment, two weeks of treatment with study drugs, and follow-up.

ELIGIBILITY:
Inclusion:

* Subjects diagnosed with nocturia, as defined by International Continence Society (i.e., the interruption of sleep one or more times at night to void), confirmed by evaluation in participating investigator's urology practice for the following characteristics: nocturia is related to overactive bladder (OAB); nightly ≥2.5 times nocturia present for at least 3 months and not considered caused by persistent or recurrent urinary tract infection; Post-Void Residual (PVR) urine volume must be <80 cc at the time of screening; did not respond well to, or unwilling to have, lifestyle modification, behavioral and conservative therapies, such as dietary changes, timed voiding, urge suppression (e.g., pelvic floor exercises [PFE] at the time of urge episodes), biofeedback, etc.
* Males or females, ≥18 years of age with Body Mass Index (BMI) <40.
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation.
* Ability to understand and sign the study Informed Consent Form (ICF), communicate with the investigators, and understand and comply with the requirements of the protocol, including completion of participation in all phases of the study.
* No current or medical history of gastrointestinal bleeding or malformation; bleeding diathesis; or restless leg syndrome.
* Not using within 4 weeks before study initiation, or anticipating the use during the study, of the following drugs: antiplatelet or anticoagulant drugs; any Selective Serotonin Re-uptake Inhibitors (SSRIs) or anti-diuretic medications; or warfarin
* Resting heart rate between 55 and 100 beats per minute, inclusive of both.

Exclusion:

* Pregnant or nursing women.
* Known presence of urinary tract infection (UTI) within 4 weeks before study initiation
* Known sleep interruptions due to sleep apnea, dyspepsia or other gastro-intestinal symptoms, seizure disorders or other neurologic symptoms
* Allergy to or intolerance of acetaminophen, ibuprofen, or any inactive component of the study drug formulations.
* A history of allergy to aspirin or other NSAIDs.
* Congenital or acquired structural abnormality of the genitourinary tract.
* Prostate cancer of any stage that has required any treatment.
* Any neurodegenerative disease (including but not limited to Parkinson's Disease, Alzheimer's Disease, Amyotrophic Lateral Sclerosis, Pick's Disease, Multi-Infarct Dementia or recent history of head trauma associated with concussion, stroke or serious cerebrovascular events) which may indicate problems in providing consistent and reliable Patient-Reported Outcomes (PRO) such as diary, Quality-of-Life, etc. required in this study.
* Uncontrolled hypertension (blood pressure >150/100 mm Hg).
* Serious medical illness, such as significant cardiac disease (e.g. symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, or New York Heart Association Class II, III or IV), severe debilitating pulmonary disease, or history of stroke (hemorrhagic or thrombotic), A-V malformation, or other cerebrovascular disease.
* Receipt of any investigational drug or participation in any clinical trial within 30 days prior to study participation.
* Use of acetaminophen, ibuprofen, acetylsalicylic acid (ASA) or any NSAID on the day of entry into the study or any anticipated use during the study. In the event of the need for any unanticipated use of such drugs during the trial, the timing and doses of such use should be carefully recorded and reported at the next visit to the clinic.
* Any medical problem requiring uninterrupted use of acetaminophen, ibuprofen, or any NSAIDs, or any other pain medication.
* Daily use of phosphodiesterase (PDE) inhibitors (such as sildenafil, tadalafil, vardenafil, avanafil, and udenafil) within 30 days prior to study or any anticipated daily use during the study. (Note: PDE inhibitors are known to have positive effect on voiding dysfunction and thus can interfere with the assessment of Paxerol [Ückert et al 2010].)
* History of polyuria or evidence of polyuria (estimation of daily production >2.5 liters of urine).
* Uncontrolled Type 1 or 2 diabetes mellitus (HbA1c >7.0%).
* Diabetes insipidus.
* Significantly impaired renal function (creatinine clearance <50 mL/min/1.73kg/m2)
* Any visual, motor or other sensory abnormality that might predispose to a fall on nocturnal arising to urinate.
* Evidence of hyponatremia at baseline.
* Any significant disease or abnormality of the neurological, visual, gastrointestinal, hepatobiliary, pulmonary, cardiovascular, genitourinary or musculoskeletal system other than those specified above that, in the opinion of the involved investigator, might compromise the ability of the prospective subject to participate in the study or that could confound interpretation of study results.
* Any abnormality on screening medical history, physical examination or clinical laboratory examination other than those specified above that, in the opinion of the involved investigator, might confound interpretation of study results.
* Subjects with known hepatitis, HIV-AIDS, or tuberculosis.
* Subjects with known dysrhythmia of any form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-01; Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Dill, Study Chair — Wellesley Pharmaceuticals
Locations (4):
- United States (4):
  - A and I Medical P.C., Brooklyn, New York
  - The Westchester Medical Group PC, Harrison, New York
  - Dr. George Klein, New York, New York
  - Washington High Urology, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee KC, Rauscher F, Kaminesky J, Ryndin I, Xie L, Zhao Y, Khusid JA, Weiss JP. Novel immediate/sustained-release formulation of acetaminophen-ibuprofen combination (Paxerol(R)) for severe nocturia associated with overactive bladder: A multi-center, randomized, double blinded, placebo-controlled, 4-arm trial. Neurourol Urodyn. 2019 Feb;38(2):740-748. doi: 10.1002/nau.23910. Epub 2018 Dec 28. PMID 30592553

RESULTS

PARTICIPANT FLOW:
Groups:
- Paxerol - Dose Level 1 325 mg Acetaminophen 150 mg Ibuprofen: Subjects are treated with the first dose level of Paxerol.
  Paxerol - Dose Level 1: Subjects are treated with the first dose level of Paxerol
- Paxerol - Dose Level 2 650 mg Acetaminophen 300 mg Ibuprofen: Subjects are treated with the second dose level of Paxerol.
  Paxerol - Dose Level 2: Subjects are treated with the second dose level of Paxerol
- Paxerol - Dose Level 3 975 mg Acetaminophen 450 mg Ibuprofen: Subjects are treated with the third dose level of Paxerol.
  Paxerol - Dose Level 3: Subjects are treated with the third dose level of Paxerol
Period: Overall Study
Arm/Group | Placebo | Paxerol - Dose Level 1 325 mg Acetaminophen 150 mg Ibuprofen | Paxerol - Dose Level 2 650 mg Acetaminophen 300 mg Ibuprofen | Paxerol - Dose Level 3 975 mg Acetaminophen 450 mg Ibuprofen
Started | 21 | 22 | 21 | 22
Completed | 19 | 22 | 20 | 21
Not Completed | 2 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: During the two week baseline period, patients completed a diary of their nightly voids. Those whose voids averaged less than 2.5 voids per night were excluded from the second two weeks of the trial. Only 86 out of the original 129 patients met this criterion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Paxerol - Dose Level 1 325 mg Acetaminophen 150 mg Ibuprofen | Paxerol - Dose Level 2 650 mg Acetaminophen 300 mg Ibuprofen | Paxerol - Dose Level 3 975 mg Acetaminophen 450 mg Ibuprofen | Total
Number analyzed (Participants) | 21 | 22 | 21 | 22 | 86
Age, Continuous [Mean (Full Range); unit: years] — The ages ranged from 34 years to 87 years old.
  years | 58.8 [34 to 87] | 60.4 [50 to 76] | 59.9 [34 to 85] | 59.9 [46 to 75] | 59.7 [34 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 7 | 18
  Male | 19 | 18 | 16 | 15 | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — The patients were found at urology clinics in the NYC area.
  participants
    United States | 21 | 22 | 21 | 22 | 86
Average nightly voids [Mean (Standard Deviation); unit: voids per night] | 3.6 (0.7) | 3.3 (1.0) | 3.9 (1.4) | 3.6 (1.0) | 3.6 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Nocturia Episodes
Description: Change in number of nocturia episodes associated with one of three dose levels of Paxerol vs. placebo is assessed during the 2-week treatment period.
Time Frame: Up to 2 weeks
Measure: Mean (Standard Deviation); unit: average nightly voids
Arm/Group | Placebo | Paxerol - Dose Level 1 325 mg Acetaminophen 150 mg Ibuprofen | Paxerol - Dose Level 2 650 mg Acetaminophen 300 mg Ibuprofen | Paxerol - Dose Level 3 975 mg Acetaminophen 450 mg Ibuprofen
Number analyzed (Participants) | 21 | 22 | 21 | 22
average nightly voids
  Baseline | 3.6 (0.7) | 3.3 (1.0) | 3.9 (1.4) | 3.6 (1.0)
  Two Weeks Using Pills | 3.2 (1.0) | 2.2 (1.0) | 2.5 (1.0) | 2.4 (1.0)
  Change of Nocturia Episodes | -0.3 (0.7) | -1.1 (0.7) | -1.4 (1.4) | -1.3 (0.8)
Statistical Analysis 1: Comparison: Placebo vs Paxerol - Dose Level 1 325 mg Acetaminophen 150 mg Ibuprofen vs Paxerol - Dose Level 2 650 mg Acetaminophen 300 mg Ibuprofen vs Paxerol - Dose Level 3 975 mg Acetaminophen 450 mg Ibuprofen; Test type: Superiority; p = 0.0017, ANOVA

2. Primary Outcome: Clinical Benefit Based on Nocturia Quality of Life (NQOL).
Description: The degree of clinical benefit, via NQOL, associated with one of three dose levels of Paxerol vs. placebo is assessed after the 2-week treatment period. This is on a scale of 0 to 100, with 0 being the best score.
Time Frame: Up to 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Paxerol - Dose Level 1 325 mg Acetaminophen 150 mg Ibuprofen | Paxerol - Dose Level 2 650 mg Acetaminophen 300 mg Ibuprofen | Paxerol - Dose Level 3 975 mg Acetaminophen 450 mg Ibuprofen
Number analyzed (Participants) | 21 | 22 | 21 | 22
score on a scale
  Baseline Quality of Life | 52.5 (15.2) | 52.3 (20.4) | 63.6 (19.6) | 59.7 (20.7)
  Two Weeks Using Pills | 42.1 (18.3) | 40.7 (21.4) | 40.5 (18.1) | 37.4 (23.4)
Statistical Analysis 1: Comparison: Placebo vs Paxerol - Dose Level 1 325 mg Acetaminophen 150 mg Ibuprofen vs Paxerol - Dose Level 2 650 mg Acetaminophen 300 mg Ibuprofen vs Paxerol - Dose Level 3 975 mg Acetaminophen 450 mg Ibuprofen; Test type: Superiority; p < .44, ANOVA

3. Secondary Outcome: Duration of First Undisturbed Sleep (DFUS)
Description: DFUS will be assessed during the 2-week treatment period with one of three dose levels of Paxerol vs. placebo
Time Frame: Up to 2 weeks
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | Paxerol - Dose Level 1 325 mg Acetaminophen 150 mg Ibuprofen | Paxerol - Dose Level 2 650 mg Acetaminophen 300 mg Ibuprofen | Paxerol - Dose Level 3 975 mg Acetaminophen 450 mg Ibuprofen
Number analyzed (Participants) | 21 | 22 | 21 | 22
Hours
  Baseline DFUS | 1.8 (0.7) | 2.2 (0.9) | 2.0 (1.1) | 2.1 (0.8)
  Two Weeks Using Pills DFUS | 2.2 (0.9) | 2.8 (1.3) | 2.7 (1.4) | 3.3 (1.5)

4. Secondary Outcome: Total Hours of Nightly Sleep
Description: The total hours of nightly sleep will be assessed during the 2-week treatment period with one of three dose levels of Paxerol vs. placebo
Time Frame: Up to 2 weeks
Measure: Mean (Standard Deviation); unit: Hours per night
Arm/Group | Placebo | Paxerol - Dose Level 1 325 mg Acetaminophen 150 mg Ibuprofen | Paxerol - Dose Level 2 650 mg Acetaminophen 300 mg Ibuprofen | Paxerol - Dose Level 3 975 mg Acetaminophen 450 mg Ibuprofen
Number analyzed (Participants) | 21 | 22 | 21 | 22
Hours per night
  Baseline Hours of Sleep | 8.5 (1.0) | 7.9 (1.0) | 8.6 (1.6) | 8.6 (1.3)
  Two Weeks Using Pills Hours of Sleep | 8.3 (1.0) | 7.7 (1.9) | 8.5 (1.4) | 8.4 (1.3)
  Change from Baseline | -0.3 (0.6) | -0.3 (0.6) | -0.2 (1.0) | -0.2 (0.6)

ADVERSE EVENTS:
Time Frame: Adverse events were tracked during the 4 week study.
Arm/Group | Placebo | Paxerol - Dose Level 1 325 mg Acetaminophen 150 mg Ibuprofen | Paxerol - Dose Level 2 650 mg Acetaminophen 300 mg Ibuprofen | Paxerol - Dose Level 3 975 mg Acetaminophen 450 mg Ibuprofen
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 4/21 | 2/22 | 3/21 | 3/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=21) | Paxerol - Dose Level 1 325 mg Acetaminophen 150 mg Ibuprofen (N=22) | Paxerol - Dose Level 2 650 mg Acetaminophen 300 mg Ibuprofen (N=21) | Paxerol - Dose Level 3 975 mg Acetaminophen 450 mg Ibuprofen (N=22)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Nausea, abdominal pain, vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Renal and Urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Glycosuria and Hematuria
Pain in flank (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Musculoskeletal and connective tissues
Hemoglobin A1c, increase (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Metabolic
Pain, chest, non-cardiac (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — General

LIMITATIONS AND CAVEATS:
None of the adverse events were considered to be drug related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT02646826/Prot_SAP_000.pdf